CLINICAL TRIAL: NCT00966420
Title: Traction Assisted Endoscopic Mucosa Resection (TAEMR)
Brief Title: Traction Assisted Polypectomy of the Intestine
Acronym: TAEMR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St John of God Hospital, Vienna (Other)
Responsible Party: Bernhard Dauser, MD, St John of God Hospital, Vienna
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SJOG-01
Record Dates: First submitted 2009-08-25; First posted 2009-08-27 (Estimated); Last update posted 2010-03-30 (Estimated); Status verified 2010-03

CONDITIONS: Colonic Polyps; Adenomatous Polyps
MeSH Terms: conditions — Colonic Polyps; Adenomatous Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- mucosa resection (Experimental)
  Interventions: Device: traction assisted endoscopic mucosa resection

INTERVENTIONS:
Device: traction assisted endoscopic mucosa resection — A haemoclip is connected to suture material and will be fixed (next) to a polyp to allow traction and lifting the lesion in order to facilitate its resection with a loop.
  Other Names: endoscopic polypectomy

SUMMARY:
The purpose of the study is to verify if the ablation of lesions (polyps, adenomas) in the large (and small) intestine can be facilitated by using a traction on the lesions.

DETAILED DESCRIPTION:
We want to facilitate the ablation of lesions (polyps, adenomas) in the large (and small) intestine by using a traction assisted technique.

The traction will be performed by using a haemoclip connected to surgical suture materials. The haemoclip will be fixed to the intestinal mucosa next to the lesion and a loop will be mounted to perform an endoscopic mucosal resection.

The aim of the study is to show the feasibility of this technique.

ELIGIBILITY:
Inclusion Criteria:

* benign lesions in the large and small intestine
* diameter of lesion smaller than 3cm

Exclusion Criteria:

* malign lesions of the large and small intestine
* diameter of lesions larger than 3cm

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-07; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
ablation of lesion in toto | 1 week after intervention

SECONDARY OUTCOMES:
complications after resection | within one week after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Dauser, MD, Principal Investigator — St John of God Hospital, Vienna
Locations (1):
- Departement of Surgery, St John of God Hospital, Vienna, Vienna, Austria